CLINICAL TRIAL: NCT07046156
Title: Evaluation of Anticholinergic Treatment Response and Predictive Factors in Pediatric Overactive Bladder
Brief Title: Treatment of Overactive Bladder With Anticholinergic Agents
Status: Active, not recruiting | Type: Observational
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Furkan Adem Canbaz, Medical doctor, Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Other Study IDs: Ivstrh - OAB
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; children; oxybutynin; propiverine; tolterodine
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — propiverine; Tolterodine Tartrate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Oxybutynin: Patients treated with oxybutynin
  Interventions: Drug: Oxybutynin Cl
- Propiverine: Patients treated with propiverine
  Interventions: Drug: propiverine
- Tolterodine: Patients treated with tolterodine
  Interventions: Drug: Tolterodine

INTERVENTIONS:
Drug: Oxybutynin Cl — Oxybutynin in a dose of 0.5 mg/kg will be used in the treatment of overactive bladder
  Groups: Oxybutynin
Drug: propiverine — Propiverine in a dose of 0.8 mg/kg will be used in the treatment of overactive bladder
  Groups: Propiverine
Drug: Tolterodine — Tolterodine in a dose of 0.1 mg/kg will be used in the treatment of overactive bladder
  Groups: Tolterodine

SUMMARY:
This study aims to evaluate the efficacy and adverse effect incidence of three different anticholinergics (oxybutinin, propiverine, and tolterodine) that are used in children with overactive bladder.

DETAILED DESCRIPTION:
A total of approximately 150 patients with overactive bladder will be evaluated retrospectively. Clinical and demographic data and voiding diaries of these patients will be evaluated. For this purpose, patients will be divided into mainly three groups according to the anticholinergic agent used.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with overactive bladder
* Patients treated with an anticholinergic

Exclusion Criteria:

* Presence of anatomical or neurological problems
* Patients with missing data

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who were treated for overactive bladder in pediatric urology clinic of Sancaktepe Sehit Prof Dr Ilhan Varank Training and Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients treated with anticholinergic | 6 months
Number of patients with drug related adverse effects | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Sancaktepe Sehit Prof dr Ilhan Varank Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ramsay S, Bolduc S. Overactive bladder in children. Can Urol Assoc J. 2017 Jan-Feb;11(1-2Suppl1):S74-S79. doi: 10.5489/cuaj.4337. PMID 28265325
- [Background] Park SJ, Pai KS, Kim JM, Park K, Kim KS, Song SH, Park S, Kim SO, Ryu DS, Baek M, Lee SD, Lee JW, Im YJ, Han SW, Chung JM, Cho MH, Ha TS, Cho WY, Suh HJ; Korean Children's Continence and Enuresis Society. Efficacy and tolerability of anticholinergics in Korean children with overactive bladder: a multicenter retrospective study. J Korean Med Sci. 2014 Nov;29(11):1550-4. doi: 10.3346/jkms.2014.29.11.1550. Epub 2014 Nov 4. PMID 25408588
- [Derived] Canbaz FA. Response to anticholinergic therapy and its predictors in pediatric overactive bladder. Eur J Pediatr. 2025 Nov 3;184(11):727. doi: 10.1007/s00431-025-06545-3. PMID 41182445